CLINICAL TRIAL: NCT02935231
Title: Proactive Minimal Cessation Advice Plus Nicotine Replacement Therapy (PMCAN) for Smoking Cessation in Smokers at Smoking Hotspots: a Pilot Randomized Controlled Trial
Brief Title: PMCAN for Smokers at Smoking Hotspots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMCANp_2016
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Smoking Cessation
Keywords: minimal cessation advice; proactive; nicotine replacement therapy; smoking hotspots
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nicotine Replacement Therapy (Experimental): This experimental group receives health warning leaflet, 1-week free nicotine replacement therapy (gum/patch), a card containing instruction and potential side effects and follow-up intervention if they have the above side effects at 3-, 7- and 10-days.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Other: Health warning leaflet
- Minimal Cessation Advice & Nicotine Replacement Therapy (Experimental): This experimental group receives brief smoking cessation advice using AWARD model with a health warning leaflet, 1-week free nicotine replacement therapy (gum/patch), a card containing instruction and potential side effects and follow-up intervention if they have the above side effects at 3-, 7- and 10-days.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Behavioral: Minimal Cessation Advice (MCA); Other: Health warning leaflet
- Minimal Cessation Advice (Experimental): This experimental group receives brief smoking cessation advice using AWARD model with a health warning leaflet.
  Interventions: Behavioral: Minimal Cessation Advice (MCA); Other: Health warning leaflet
- Control (Active Comparator): This control group receives a health warning leaflet.
  Interventions: Other: Health warning leaflet

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (NRT) — 1-week free NRT (gum/patch) plus a card containing instruction and potential side effects.
  Other Names: NRT
  Arms: Minimal Cessation Advice & Nicotine Replacement Therapy; Nicotine Replacement Therapy
Behavioral: Minimal Cessation Advice (MCA) — Brief smoking cessation advice using AWARD model. AWARD: (1) Ask smoking habit; (2) Warn about smoking risk; (3) Advice to quit as soon as possible; (4) Refer to smoking cessation service; and (5) Do-it-again: if relapse/fail.
  Other Names: MCA
  Arms: Minimal Cessation Advice; Minimal Cessation Advice & Nicotine Replacement Therapy
Other: Health warning leaflet — An A4 double-side color leaflet containing shocking pictures of diseases associated with smoking.

SUMMARY:
Background: Many smokers cannot quit due to nicotine withdrawal symptoms, which peak at the first week of abstinence. Proactive recruitment of smokers is needed as most smokers do not seek smoking cessation (SC) services. A smoking hotspot (SH) is defined as a public outdoor place where smokers stop/linger and smoke. We aim to include a reasonably "representative" or unbiased sample of SH at different locations from all 3 regions of Hong Kong. We will randomly select 6 eligible SH (2 in each regions) from the 15 hotspots in our previous community trial.

Methods: Two trained SC ambassadors (student helpers) and one supervisor (experienced research assistant) will be deployed for each session of intervention at a SH. Potential subjects will be approached using the "a-foot-into-the-door" method in which SC ambassador will ask if smoker would like to reduce/quit smoking and receive SC intervention or advices. Smokers will be assessed for eligibility and informed written consent will be sought. Subjects will complete a brief self-administered questionnaire (baseline) using tablet. To reduce later hang-ups of telephone interventions or surveys, SC ambassador will save contact number of the trial into subjects' mobile phones.

Discussion: The findings will provide much needed and original evidence to support a main RCT on these new, proactive, simple and low-cost interventions for improving current SC services and policy for smokers who do not actively seek help from SC services in Hong Kong and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Adult smokers aged 18+ who smoke cigarettes daily.
* Exhaled carbon monoxide (CO) level of 4ppm or above.
* Hong Kong residents able to read and communicate in Chinese (Cantonese or Putonghua)

Exclusion Criteria:

* Smokers who have contraindication for NRT use: severe angina, arrhythmia, myocardia infraction, pregnancy (or intended to become pregnant <6 months) or breastfeeding.
* Smokers who have psychiatric/psychological diseases or regular psychotropic medications
* Smokers who are using SC medication, NRT, other SC services or projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Exhaled CO validated abstinence | 3 month

SECONDARY OUTCOMES:
Self-reported past 7-day point prevalence abstinence | 3 month
Nicotine Replacement Therapy use | 3 month
Smoking cessation service use | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping WANG, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided